CLINICAL TRIAL: NCT04572334
Title: Repeatability of Post-operative Refraction in Patients With a Novel CE Marked Monofocal Intraocular Lens
Brief Title: Eyhance Autorefraction Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of the Ophthalmology Department, and Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Eyhance Autorefraction study
Record Dates: First submitted 2020-09-30; First posted 2020-10-01 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Cataract Senile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual acuity and refractive outcome for Tecnis Eyhance (Other): Evaluation the comparability and reproducibility of different refraction methods in patients implanted with Eyhance lens
  Interventions: Other: Auto and Subjective Refraction
- visual acuity and refractive outcome for Tecnis ZCB00 (Other): Evaluation the comparability and reproducibility of different refraction methods in patients implanted with ZCB00 lens
  Interventions: Other: Auto and Subjective Refraction

INTERVENTIONS:
Other: Auto and Subjective Refraction — All patients will be measured with three autorefractometers and two independent observes will perform subjective refraction

SUMMARY:
Since 2018, the Tecnis Eyhance ICB00 lens (Johnson&Johnson Vision, AMO Germany GmbH) was introduced, which is a monofocal IOL which has the ability of extended depth of focus improving intermediate vision without the photic phenomena specific for the multifocal IOLs. The Tecnis Eyhance ICB00 is one of our standard IOL, routinely used in our clinic. There is no single outcome measurement that can be thought of as summarizing the efficacy of an IOL, nevertheless visual acuity and refractive outcome are the most important parameters for evaluation. Aim of this study is to determine the comparability and reproducibility of different refraction methods in patients implanted with Eyhance lens and compare the outcomes with ZCB00 lens.

DETAILED DESCRIPTION:
This a prospective observational study that would include pseudophakic patients that have undergone cataract surgery 2 to 12 months prior. A written informed consent will be obtained from each patient. Patients with ICB00 or ZCB00 implanted lenses will be included.

Autorefraction measurements will be performed consecutively, each patient will be measured three times with each device. Two independent observers will perform subjective refraction and will be masked to the autorefraction outcome.

We would like to include 50 eyes with ICB00 and 50 eyes with ZCB00 lens implanted. For the estimation of sample size, we used data from Wang et al. (Wang L, Misra M, Palikaris IG, Koch DD. J Cataract Refract Surg 2002; 28: 276-282) that compared the refractive outcome of pseudophakic eyes and determined a mean spherical equivalent of -0.76 + 0.96 D for group I and -0.44 + 1.13 for group II, thus leading to an effect size of 0.2. The effect size was used for ANOVA test for repeated measurements within factor, with alpha < 0.05, power of 80% and a correlation of 0.5 between the two groups gave us an estimated of sample size of 42 patient. To allow patient drop out a number of 50 eyes will be included per lens group (in total 100 eyes).

When different lenses are implanted (one eye received ZCB00 and the other Eyhance), than both eyes of the patient will be included.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or above
* Operated age-related cataract (pseudophakic patient)
* Tecnis Eyhance ICB00 or Tecnis ZCB00 IOL implanted within 2 to 12 months prior to study related examination

Exclusion Criteria:

* Intra- or Postoperative complication
* patients with severe corneal pathology, severe macular degeneration, severe diabetic retinopathy, etc. that would significantly influence visual outcome
* nystagmus or pathologies that would affect patient fixation
* pregnancy- for women in reproductive age a pregnancy test will be performed.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of different refraction methods | 2-12 months

SECONDARY OUTCOMES:
Comparability between the devices (autorefractometers) | 2-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No